CLINICAL TRIAL: NCT03081650
Title: The Efficacy of the AIRVO Warm Humidifier as an Add on to Oxygen Therapy as Well as Stand-alone Therapy in Patients With Respiratory Insufficiency
Brief Title: The Efficacy of the AIRVO Warm Humidifier as an Add on to Oxygen Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lutheran Hospital, Indiana (Other)
Collaborators: Fisher and Paykel Healthcare (Industry)
Responsible Party: Principal Investigator, Eustice Fernandes MD, Principal Investigator, Lutheran Hospital, Indiana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-454
Record Dates: First submitted 2017-02-22; First posted 2017-03-16 (Actual); Last update posted 2017-03-16 (Actual); Status verified 2017-02

CONDITIONS: COPD; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The study will be conducted as an open label, non-randomized trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective Open label (Experimental): All of the patients that will be Selected to participate in the study will be given an AIRVO humidifier by the study sponsor. Patients will be connected to and instructed in the use of the AIRVO. The total flow will be set at 20-25 L/min, exact flow rate will be dependent on the patient's preference. Optiflow oxygen catheter will be used to ensure against unpleasant sensation due to high flow and to avoid push back in the system.
  When acceptable flow rated has been established, it is recorded in the patient's folder. The patients is then instructed to use the AIRVO for a minimum eight (8) hour period, preferably at night. Using the humidifier for a longer period of time is allowed. The total number of hours the humidifier was operational will be recorded at the end of the study
  Interventions: Device: Airvo Humidifier

INTERVENTIONS:
Device: Airvo Humidifier

SUMMARY:
The primary purpose of this study is to show whether at home usage of the AIRVO warm humidifier can potentially reduce the number of exacerbations in patients with significant respiratory insufficiency. Eligible participants of the study must have a diagnosis of chronic obstructive pulmonary disease (COPD) stage II-IV..

DETAILED DESCRIPTION:
SPECIFIC AIMS/OBJECTIVES To determine whether the patients with chronic respiratory sufficiency can benefit from the AIRVO warm humidifier by decreasing the number of exacerbations. Furthermore, to determine the efficacy of warm humidification oxygen therapy compared to dry oxygen therapy, in short-term and long-term treatment of patients with stage II-IV COPD.

Primary Objective:

To observer and compare the exacerbation frequency between the warm humidification oxygen therapy group and dry oxygen therapy group.

Secondary Objective:

Compare the number of exacerbation days, median time to first exacerbation, hospital readmissions, and antibiotic use pertaining to respiratory infections with the baseline values. Evaluate and compare the quality of life to the baseline measurements.

STUDY OVERVIEW

Methods:

The study will be conducted as an open label, non-randomized trial. Patients will be assigned to AIRVO humidification if they meet all of the inclusion/exclusion criteria of the study. All of the study participants will have the AIRVO warm humidifier installed at their home as a stand alone unit or in addition to their current LTOT therapy. For the patients that are already on LTOT, the oxygen flow setting will be increased to 20-25 l/min, to the optimum flow by taking in consideration the patient's preference.

Data:

Data to be collected includes exacerbation frequency, number of exacerbation days, and time to first exacerbation, pulmonary functions test, antibiotic usage and Quality of Life assessment.

Description of AIRVO:

The AIRVO is for the treatment of spontaneously breathing patients who would benefit from receiving high flow warmed and humidified respiratory gases. The AIRVO humidifier has adjustable flow setting for delivery of fully saturated breathing gases at 37°C, 100% humidity.

Flow rates on the humidifier are adjustable between 10 and 60 L/min for this specific population (general is 2 -60 L/min). AIRVO humidifier is intended to be used in combination with medical oxygen supply. When coupled to a medical oxygen supply, the regulation of oxygen concentration is ensured, allowing for treatment of COPD patients with greater oxygen flow without risking an increased accumulation of carbon dioxide. The mixed gases, atmospheric air and with medical oxygen, pass through a humidification chamber with sterile water for humidification and heating. Breathing tubes are equipped with spiral wire, this aids with heating and ensures the uniform temperature and humidity is maintained. The air is supplied to the patients at 37°C, 100% humidity. [16]

Treatment groups:

ARIVO:

All of the patients that will be Selected to participate in the study will be given an AIRVO humidifier by the study sponsor. Patients will be connected to and instructed in the use of the AIRVO. The total flow will be set at 20-25 L/min, exact flow rate will be dependent on the patient's preference. Optiflow oxygen catheter will be used to ensure against unpleasant sensation due to high flow and to avoid push back in the system.

When acceptable flow rate has been established, it is recorded in the patient's folder. The patients is then instructed to use the AIRVO for a minimum eight (8) hour period, preferably at night. Using the humidifier for a longer period of time is allowed. The total number of hours the humidifier was operational will be recorded at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

Have stage II-IV COPD diagnosis Understand and accept oral and written information in English Be capable of handling the AIRVO warm humidifier after instruction >18years of age

Exclusion Criteria:

* Comorbidity (known malignant disease, terminal illness, dementia, uncontrolled mental illness)
* Bronchiectasis without simultaneous COPD diagnosis
* Treatment with BiPAP in the home
* Affected level of consciousness
* Smoking status change during study period
* Inability to provided signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-08-16 (Actual); Primary Completion 2017-08-16 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
The change in number of hospitalizations warm humidification oxygen therapy and dry oxygen therapy. | baseline, 12 months
  The change in number of hospitalizations compared to baseline data at 12 months.
Change in the number of courses of antibiotic therapy compared to baseline data at 12 months | baseline, 12 months
Change in the number of courses of corticosteroid therapy compared to baseline data at 12 months. | baseline, 12 months
Change in the number of COPD medication therapy changes compared to baseline at 12 months. | baseline, 12 months

SECONDARY OUTCOMES:
Change in Spirometry measured pulmonary function between humidification oxygen therapy and dry oxygen therapy at baseline, and 12 months. | baseline, 12 months
  Change in Spirometry measured Pulmonary function test ( FEV1 and FEV1/FVC Forced vital capacity 1 (FEV1)- Volume forced expiration at 1.0, second in liters Forced Vital capacity - (FVC) Total amount of air in liters measured during a forced expiratory breath and peak expiratory flow) compared to baseline at 12 months
The change in distance walked during a 6 minute walk test between humidification oxygen therapy and dry oxygen therapy at baseline, and 12 months. | baseline, 12 months
  Change in 6 minute walk test (the distance walked in feet over a 6 minute period) compared to baseline at 12 months
The change in the quality of life scores as measured by the Ferrans and Powers quality of life Index Pulmonary version III between humidification oxygen therapy and dry oxygen therapy at baseline, and 12 months. | baseline, 12 months
  The change in the QOL measurements, (Ferrans and Powers Quality of Life Index Pulmonary Version -III, A two part 1 through 6 scaled survey, 1 very dissatisfied & 6 Very satisfied. The first part focuses on how satisfied you are with the area of your life and the second on how important that area of your life is to you. Each section is comprised of 36 questions.) compared to baseline at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Eustace Fernandes, MD, Principal Investigator — Lutheran hospital
Locations (1):
- Lutheran hospital, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ringbaek TJ, Viskum K, Lange P. Does long-term oxygen therapy reduce hospitalisation in hypoxaemic chronic obstructive pulmonary disease? Eur Respir J. 2002 Jul;20(1):38-42. doi: 10.1183/09031936.02.00284202. PMID 12166578
- [Background] Continuous or nocturnal oxygen therapy in hypoxemic chronic obstructive lung disease: a clinical trial. Nocturnal Oxygen Therapy Trial Group. Ann Intern Med. 1980 Sep;93(3):391-8. doi: 10.7326/0003-4819-93-3-391. PMID 6776858
- [Background] Golar SD, Sutherland LL, Ford GT. Multipatient use of prefilled disposable oxygen humidifiers for up to 30 days: patient safety and cost analysis. Respir Care. 1993 Apr;38(4):343-7. PMID 10145893
- [Background] Yamashita K, Nishiyama T, Yokoyama T, Abe H, Manabe M. A comparison of the rate of bacterial contamination for prefilled disposable and reusable oxygen humidifiers. J Crit Care. 2005 Jun;20(2):172-5; discussion 175. doi: 10.1016/j.jcrc.2005.01.002. PMID 16139158
- [Background] Loew DA, Klein SR, Chalon J. Volume-controlled relative humidity using a constant-temperature water vaporizer. Anesthesiology. 1972 Feb;36(2):181-4. doi: 10.1097/00000542-197202000-00024. No abstract available. PMID 5059111
- [Background] Salah B, Dinh Xuan AT, Fouilladieu JL, Lockhart A, Regnard J. Nasal mucociliary transport in healthy subjects is slower when breathing dry air. Eur Respir J. 1988 Oct;1(9):852-5. PMID 3229484
- [Background] Miyamoto K, Nishimura M. Nasal dryness discomfort in individuals receiving dry oxygen via nasal cannula. Respir Care. 2008 Apr;53(4):503-4. No abstract available. PMID 18397537
- [Background] Franchini ML, Athanazio R, Amato-Lourenco LF, Carreirao-Neto W, Saldiva PH, Lorenzi-Filho G, Rubin BK, Nakagawa NK. Oxygen With Cold Bubble Humidification Is No Better Than Dry Oxygen in Preventing Mucus Dehydration, Decreased Mucociliary Clearance, and Decline in Pulmonary Function. Chest. 2016 Aug;150(2):407-14. doi: 10.1016/j.chest.2016.03.035. Epub 2016 Apr 2. PMID 27048871
- [Background] Rea H, McAuley S, Jayaram L, Garrett J, Hockey H, Storey L, O'Donnell G, Haru L, Payton M, O'Donnell K. The clinical utility of long-term humidification therapy in chronic airway disease. Respir Med. 2010 Apr;104(4):525-33. doi: 10.1016/j.rmed.2009.12.016. Epub 2010 Feb 9. PMID 20144858
- [Background] Wier LM, Elixhauser A, Pfuntner A, Au DH. Overview of Hospitalizations among Patients with COPD, 2008. 2011 Feb. In: Healthcare Cost and Utilization Project (HCUP) Statistical Briefs [Internet]. Rockville (MD): Agency for Healthcare Research and Quality (US); 2006 Feb-. Statistical Brief #106. Available from http://www.ncbi.nlm.nih.gov/books/NBK53969/ PMID 21510031
- See also: What is COPD? National Heart Lung and Blood Institute: Diseases and Conditions Index. June 2010. — http://www.nhlbi.nih.gov/health/dci/Diseases/Copd/copd_WhatIs.html.